CLINICAL TRIAL: NCT01314300
Title: VERSATIS - Efficacy and Safety of Lidocaine 5% Plasters (Versatis® 5%) in Child, Adolescents and Young Adults With Neuropathic Pains or Vasoocclusive Sickle Cell Crisis Pains
Brief Title: Lidocaine 5% Plasters (Versatis® 5%) in Pediatric Neuropathic Pains and Vasoocclusive Sickle Cell Crisis Pains
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VERSATIS
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Neuropathic Pains; Vasoocclusive Sickle Cell Crises Pains
Keywords: Child, adolescent, young adult; Plaster; Lidocaine
MeSH Terms: conditions — Neuralgia | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Efficacy of Lidocaine 5% plaster (Experimental): Treatment of pain by Lidocaine 5% plaster
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 5% plaster
  Other Names: Versatis® 5%

SUMMARY:
Lidocaine 5% plaster (VERSATIS® 5%) showed its efficacy and safety in the post-herpetic zoster adult pains. This treatment is recommended in first intention in adult neuropathic pains with allodynia.

The purpose of this study is to assess efficacy and safety of lidocaine 5% plaster (VERSATIS® 5%) in the pediatric neuropathic pains and vasoocclusive sickle cell crises pains.

DETAILED DESCRIPTION:
Pediatric neuropathic pain are infrequent. It's difficult to estimate the prevalence. It may result from several causes : infectious (post-herpetic neuropathy), traumatic (tumor or Positional)or toxic (chemotherapy or radiotherapy). They are often associated with malignant pediatric disease.

These pains are spontaneous, continuous or intermittent, as type of burns or electric shocks or abnormal skin sensation (hyperesthesia or allodynia). Treatment is the same as in adults: antiepileptic or neuroleptics, sometimes associated with analgesic (level 2 or 3).

Lidocaine 5% plaster are used in adults as first line of treatment to reduce post-herpetic neuropathic pain, especially in cases of mechanical allodynia. These plasters are indicated for the symptomatic treatment of post-herpetic neuropathic pain.

Each plaster contains 700 mg of lidocaine. It must be applied on the painful area once daily for a maximum period of 12 hours per 24 hours.

The primary endpoint is to evaluate the efficacy of lidocaine 5% plaster (VERSATIS 5%) after 12 hours on reducing of pure or mixed neuropathic pain and on reducing of vasoocclusive sickle cell pain, localized, superficial, in child, adolescent and young adult.

The secondary endpoint are:

1. to evaluate the efficacy of lidocaine 5% plaster (VERSATIS 5%) after 6 hours on reducing of pure or mixed neuropathic pain and on reducing of vasoocclusive sickle cell pain, localized, superficial, in child, adolescent and young adult.
2. to evaluate safety of lidocaine 5% plaster (VERSATIS® 5%) in these same indications.

ELIGIBILITY:
Inclusion Criteria:

* 6 years <= Age <= 21 years
* With:

  * Pure or mixed, localized, superficial neuropathic pains for which the neuropathic pain score DN4 is greater than or equal to 4
  * Or localized, superficial sickle cell crisis pains Insufficiently relieved by commonly used therapeutic (analgesic level II or III and / or antiepileptic drugs, and / or neuroleptics) - GCS > 12
* Covered by a medical insurance
* Signed written informed consent form(for minors unemancipated, permission will be given by holders of parental authority)

Exclusion Criteria:

* Clinical condition not permitting data reporting (impaired consciousness)
* Painful area with an surface greater than:

  * 150 cm² for a patient with total body surface area < 1 m²
  * 300 cm² for a patient with 1 m² < total body surface area < 1.5 m²
  * 450 cm² for a patient with total body surface area > 1.5 m²
* Existence of a statement for the use of lidocaine 5% (VERSATIS® 5%) plaster as defined in the summary of product characteristics, as:

  * known hypersensitivity to the active substance or excipients
  * known hypersensitivity to other local anesthetics such as amide (eg bupivacaine, etidocaine, mepivacaine and prilocaine)
  * inflammatory or injured skin (active lesions of herpes zoster, dermatitis or wounds)
* Severe cardiac insufficiency
* Severe renal insufficiency
* Severe hepatic insufficiency
* Patient receiving anti-arrhythmic class I or other local anesthetics.
* Pregnant or lactating female or female of child-bearing potential not employing adequate contraception
* Patient included in another clinical trial on the management of pain

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Lidocaine 5% plaster efficacy between t0 and t12 | 12 hours
  Rate of patients with a decrease of at least 2 points in pain score (at least 2 of 3 consecutive days) measured by self-assessment on a visual analogue scale (VAS) graded from 0 to 10 (0 = absence pain and 10 = maximal pain ), between start of treatment(t0) and a measure carried out 12 hours later (t12).

SECONDARY OUTCOMES:
Lidocaine 5% plaster efficacy between t0 and t6 | 6 hours
  Rate of patients with a decrease of at least 2 points in pain score (at least 2 of 3 consecutive days) measured by self-assessment on a visual analogue scale (VAS) graded from 0 to 10 (0 = absence pain and 10 = maximal pain ), between start of treatment(t0) and a measure carried out 6 hours later (t6).
Lidocaine 5% plaster safety | 72 hours
  Rate of patients with local and/or general adverse event as graded using NCI-CTCAE V4.0

CONTACTS AND LOCATIONS:
Overall Officials: Perrine MAREC-BERARD, M.D., Principal Investigator — IHOP
Locations (2):
- France (2):
  - IHOP, Lyon
  - Centre Médico-chirurgical de Réadaptation des Massues, Lyon

REFERENCES:
- [Result] Walker SM. Pain in children: recent advances and ongoing challenges. Br J Anaesth. 2008 Jul;101(1):101-10. doi: 10.1093/bja/aen097. Epub 2008 Apr 21. PMID 18430745
- [Result] Walco GA, Dworkin RH, Krane EJ, LeBel AA, Treede RD. Neuropathic pain in children: Special considerations. Mayo Clin Proc. 2010 Mar;85(3 Suppl):S33-41. doi: 10.4065/mcp.2009.0647. PMID 20194147
- [Result] Garnock-Jones KP, Keating GM. Lidocaine 5% medicated plaster: a review of its use in postherpetic neuralgia. Drugs. 2009 Oct 22;69(15):2149-65. doi: 10.2165/11203220-000000000-00000. PMID 19791831
- [Result] Rowbotham MC, Davies PS, Verkempinck C, Galer BS. Lidocaine patch: double-blind controlled study of a new treatment method for post-herpetic neuralgia. Pain. 1996 Apr;65(1):39-44. doi: 10.1016/0304-3959(95)00146-8. PMID 8826488